CLINICAL TRIAL: NCT05565807
Title: A Phase Ib/IIa, Open-Label, Dose-Escalation and Extension Study to Evaluate the Safety and Efficacy of An Anti-CD38 Antibody Drug Conjugate (STI-6129) in Patients With Relapsed or Refractory Multiple Myeloma
Brief Title: Safety and Efficacy Study of An Anti-CD38 Antibody Drug Conjugate in Relapsed or Refractory Multiple Myeloma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Zhejiang ACEA Pharmaceutical Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 38ADC-RRMM-C101
Record Dates: First submitted 2022-09-27; First posted 2022-10-04 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Relapsed or Refractory Multiple Myeloma
MeSH Terms: conditions — Recurrence; Multiple Myeloma

STUDY DESIGN:
Intervention Model Description: To determine DLT and RP2D, the design uses a accelerated titration design and a 3+3 design for the dose-escalation stage.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- STI-6129 (Experimental): Nine dosing cohorts will be evaluated: 0.25 mg/kg，0.50 mg/kg，0.67 mg/kg, 0.88 mg/kg, 1.18 mg/kg, 1.56 mg/kg, 2.08 mg/kg, 2.77 mg/kg, 3.68 mg/kg where STI-6129 will be intravenously administered once as part of a 4-week treatment cycle.
  Interventions: Biological: STI-6129

INTERVENTIONS:
Biological: STI-6129 — Anti-CD38 A2 human antibody drug conjugate (ADC) containing an antibody covalently bound to a duostatin tubulin inhibitor.

SUMMARY:
This is a phase Ib/IIa, open-label, dose-escalation, and extension study to evaluate the safety and efficacy of an anti-CD38 antibody drug conjugate (STI-6129) in patients with relapsed or refractory multiple myeloma.

DETAILED DESCRIPTION:
This is a phase Ib/IIa, open-label, dose-escalation, and extension study to evaluate the safety and efficacy of an anti-CD38 antibody drug conjugate (STI-6129) in patients with relapsed or refractory multiple myeloma.

The study is designed to identify the recommended phase 2 dose (RP2D) of STI-6129 by assessing the safety, preliminary efficacy and pharmacokinetics using a accelerated titration design and a conventional 3+3 study design for dose escalation in stage one and then the second stage will be an expansion study to assess preliminary efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old, regardless of gender.
2. Previously treated with at least three drugs (including PI, IMiD, and anti-CD38 antibody), and relapsed/refractory after the most recent anti-MM therapy.
3. Diagnosis of MM according to IMWG criteria with measurable lesions, meeting at least 1 of the following criteria:

   * Serum M protein ≥ 0.5g/dL (≥ 5 g/L); or
   * Urine M protein ≥ 200mg/24 hours; or
   * When the serum free light chain (FLC) ratio is abnormal, the affected FLC level is ≥10mg/dL (≥100 mg/L) (the normal FLC ratio is 0.26 to 1.65).
4. ECOG performance status score is 0, 1, or 2.
5. Willing and able to comply with the study schedule and all other study protocol requirements.
6. Women of childbearing potential (WOCBP) (infertile women are defined as sexually mature females who had undergone a hysterectomy or bilateral oophorectomy or bilateral salpingectomy or bilateral tubal ligation/closure, or who are infertile due to a congenital or acquired condition or spontaneously menopausal for ≥ 12 months) must have a negative blood pregnancy test during the screening. Female subjects of childbearing potential and male subjects with fertility must use a highly effective method of contraception from screening to 6 months after the last treatment.

Exclusion Criteria:

1. Known hypersensitivity to any of the ingredients of this product.
2. Diagnosis of active plasma cell leukemia.
3. Diagnosis of systemic light chain amyloidosis.
4. MM involving the central nervous system.
5. Has POEMS syndrome.
6. There is spinal cord compression associated with MM.
7. Needs to take concomitant drugs with a strong inhibitory effect or a strong induction effect on CYP3A4.
8. Had received plasma exchange therapy within 28 days before the first administration of the study drug.
9. Had received the following anti-tumor treatments before the first administration of the study drug: monoclonal antibody or cytotoxic drug or radiotherapy within 28 days; immunoregulator, targeted therapy or epigenetic therapy or investigational medical product or invasive investigational medical device or other anti-myeloma therapy within 28 days or 5 half-lives (whichever is shorter); proteasome inhibitor or anti-tumor traditional Chinese medicine treatment or corticosteroids with a cumulative dose of more than 140 mg prednisone (or equivalent) or a single dose of more than 40 mg/day dexamethasone (or equivalent) within 14 days.
10. Had received CAR-T therapy or allogeneic hematopoietic stem cell transplantation therapy within 6 months before the first administration of the study drug, or have a concomitant disease of active graft-versus-host disease (GvHD) at screening.
11. Had received autologous hematopoietic stem cell transplantation within 12 weeks before the first administration of the study drug.
12. Had undergone major surgery or eye surgery within 28 days before the first administration of the study drug.
13. Other malignant diseases within 3 years before the first administration of the study drug.
14. History of grade ≥3 (muscle paralysis, eyelid disease, glaucoma requiring drug control, tearing eyes), or grade ≥2 any other ocular disease (as judged by NCI-CTCAE version 5.0) at screening.
15. Has ≥ Grade 3 neuropathy or Grade 2 neuropathy with associated pain.
16. The toxicity caused by the previous anti-tumor treatment did not subside to ≤ grade 1.
17. Has the following hematological test results within 7 days before the first administration of the study drug:

    1. Hemoglobin <80g/L
    2. Platelet count <50×10^9/L
    3. Absolute neutrophil count <1.0×10^9/L
18. Has the following blood chemistry test results within 7 days before the first administration of the study drug:

    1. Estimated creatinine clearance <30mL/min.
    2. AST or ALT>3×upper limit of normal (ULN) or serum total bilirubin> 1.5×ULN.
19. Severe or uncontrolled cardiovascular and cerebrovascular diseases requiring treatment, including:

    1. New York Heart Association class>2;
    2. Unstable angina pectoris that cannot be controlled by drugs;
    3. Myocardial infarction occurred within 6 months before the first administration of the study drug;
    4. Poorly controlled arrhythmias;
    5. 12-lead ECG QTcF>470msec;
    6. Left ventricular ejection fraction <40%;
    7. Poorly controlled hypertension ;
    8. Stroke, cerebrovascular accident, or transient ischemic attack occurred within 6 months before the first administration of the study drug.
20. Meets any of the following criteria:

    1. Known chronic obstructive pulmonary disease (COPD) and forced expiratory volume in 1 second (FEV1) <50% of predicted normal;
    2. Known moderate or severe persistent asthma, or a history of asthma within the past 2 years, or current uncontrolled asthma of any classification;
    3. with interstitial lung disease requiring corticosteroid therapy, drug-induced interstitial lung disease, a history of radiation pneumonitis, orclinically active interstitial lung disease suggested by any current evidence before the first administration of the study drug.
21. Has an active bacterial, viral, or fungal infection or needs for intravenous antibiotic administration (IV) within 72 hours before the first administration of the study drug.
22. Active or uncontrolled HBV , HCV , HIV positive.
23. Is currently pregnant or breast feeding.
24. Has any active severe mental illness, medical illness, or other symptoms/conditions that may affect treatment, compliance, or the ability to provide informed consent, as determined by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2023-02-09 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-02-19 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events（AEs） | Up to 2 years
  Assessing the incidence of adverse events (AEs) using the Common Terminology Criteria for Adverse Events (CTCAE Version 5).
Overall response rate（ORR） | Up to 2 years
  ORR assessed by the modified IMWG response criteria.

SECONDARY OUTCOMES:
Plasma concentration of the total anti-CD38 antibody | Up to 2 years
  Determine plasma levels of the total antibody.
Plasma concentration of conjugated toxin | Up to 2 years
  Determine plasma levels of conjugated toxin (STI 6129).
Plasma concentration of the free toxin | Up to 2 years
  Determine plasma levels of the free toxin (duostatin 5.2).
Recommended Phase 2 dose (RP2D) | Up to 2 years
  Determined according to the phase 1b.
Progression-Free Survival | Up to 2 years
  PFS is the period from patient enrollment until PD or death.
Overall Survival (OS) | Up to 2 years
  OS is the period from enrollment until death from any cause.
Time To First Response（TTR） | Up to 2 years
  TTR is the period from the date of patient registration to the date of first response.
Duration of Response (DOR) | Up to 2 years
  DOR is the period from the first documentation of response (CR or PR) to the first documentation of PD.
Clinical Benefit Rate (CBR) | Up to 2 years
  CBR is the percentage of participants achieving a CR or PR at any time during the study or maintaining stable disease for at least 4 weeks from the first dose of study intervention.

CONTACTS AND LOCATIONS:
Overall Officials: jie jin, doctor, Principal Investigator — Zhejiang University; juan li, doctor, Principal Investigator — First Affiliated Hospital, Sun Yat-Sen University
Locations (4):
- China (4):
  - Beijing Chao-Yang Hospital，Capital Medicine University, Beijing, Beijing Municipality
  - Peking university Third hospital, Beijing, Beijing Municipality
  - The first affiliated hospital ,Sun Yat-sen University, Guangzhou, Guangdong
  - The First Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang